CLINICAL TRIAL: NCT02736968
Title: Phase IIa Randomized, Single-Blinded, Placebo-Controlled Clinical Trial of the Reprofiled Drug Auranofin for GI Protozoa
Brief Title: Auranofin for Giardia Protozoa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0015
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2020-04-21

CONDITIONS: Amoebic Dysentery; Giardiasis
Keywords: Amebiasis; Auranofin; GI Protozoa; Giardiasis; Placebo-Controlled; Reprofiled Drug; Single-Blind
MeSH Terms: conditions — Dysentery, Amebic; Giardiasis; Amebiasis | interventions — Auranofin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- E. histolytica- Active (Experimental): N=34, 6mg auranofin daily x 7 days
  Interventions: Drug: Auranofin
- E. histolytica- Placebo (Placebo Comparator): N=34, 6mg placebo daily x 7 days
  Interventions: Other: Placebo
- Giardia- Active (Experimental): N=34, 6mg auranofin daily x 5 days
  Interventions: Drug: Auranofin
- Giardia- Placebo (Placebo Comparator): N=34, 6mg placebo daily x 5 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Auranofin — Auranofin is a gold-containing chemical salt available as 3mg capsules
  Arms: E. histolytica- Active; Giardia- Active
Other: Placebo — Placebo
  Arms: E. histolytica- Placebo; Giardia- Placebo

SUMMARY:
This is a phase IIa, randomized, placebo-controlled, single-blinded superiority treatment study in males and non-pregnant females, 18 to 65 years of age who are in good health. This study is designed to compare placebo to once daily doses of 6mg auranofin for adults with amebiasis or giardiasis. A sample size of 68 subjects enrolled with amebiasis (34 per arm) and 68 with giardiasis (34 per arm); Power based on 60 subjects with amebiasis and 60 with giardiasis completing the study.Eligible subjects will be randomly assigned to a treatment group with auranofin (6 mg orally once daily for 5 days for giardiasis or 7 days for amebiasis) compared to a placebo group receiving similar but not identical placebo capsules. Projected duration of subject participation will be approximately 30 days of face to face visits, including the pre-enrollment screening period of up to 4 days. It is anticipated that it will take approximately 3.5 years to finish the study. Primary objectives are: 1) to compare the proportion of subjects with stools positive by rapid Enzyme Immunoassay (EIA) and positive antigen detection EIA for E. histolytica at enrollment with resolution of diarrhea (less than 3 loose stools/24 hrs) by Day 7 for E. histolytica infections. 2) to compare the proportion of subjects with stools positive by rapid EIA and positive antigen detection EIA for Giardia at enrollment with resolution of diarrhea (less than 3 loose stools/24 hrs) by Day 5 for Giardia infections.

DETAILED DESCRIPTION:
This is a phase IIa, randomized, placebo-controlled, single-blinded superiority treatment study in males and non-pregnant females, 18 to 65 years of age who are in good health. This study is designed to compare placebo to once daily doses of 6mg auranofin for adults with amebiasis or giardiasis. A sample size of 68 subjects enrolled with amebiasis (34 per arm) and 68 with giardiasis (34 per arm); Power based on 60 subjects with amebiasis and 60 with giardiasis completing the study. Eligible subjects will be randomly assigned to a treatment group with auranofin (6 mg orally once daily for 5 days for giardiasis or 7 days for amebiasis) compared to a placebo group receiving similar but not identical placebo capsules. Projected duration of subject participation will be approximately 30 days of face to face visits, including the pre-enrollment screening period of up to 4 days. It is anticipated that it will take approximately 3.5 years to finish the study. Primary objectives are: 1) to compare the proportion of subjects with stools positive by rapid Enzyme Immunoassay (EIA) and positive antigen detection EIA for E. histolytica at enrollment with resolution of diarrhea (less than 3 loose stools/24 hrs) by Day 7 for E. histolytica infections. 2) to compare the proportion of subjects with stools positive by rapid EIA and positive antigen detection EIA for Giardia at enrollment with resolution of diarrhea (less than 3 loose stools/24 hrs) by Day 5 for Giardia infections. Secondary objectives for E. histolytica infections are: 1) to compare the proportion of subjects with stools positive by rapid EIA and positive antigen detection EIA for E. histolytica and trophozoites on smear at enrollment with parasitological response (no detection of trophozoites of E. histolytica on microscopic exam) by Day 7; 2) to compare the proportion of subjects with stools positive rapid EIA and positive antigen detection EIA for E. histolytica and trophozoites on smear at enrollment with parasitological response (no detection of trophozoites on microscopic exam or negative antigen detection) by Days 3 and 5; 3) to compare the rate of decrease of trophozoites/cyst load by Quantitative Polymerase Chain Reaction (qPCR) in stools by Days 3, 5, and 7; 4) to compare the proportion of subjects with negative stool antigen tests by days 3, 5, 7, and 14; 5) to compare the proportion of subjects with sustained cure (no detection of trophozoites by microscopic exam) at 14 and 28 days; 6) to compare the proportion of subjects with relapse (same strain) or re-infection (new strain) with positive stools at 14 and 28 days by genotyping the initial vs. subsequent strain; 7) to compare the time to resolution of diarrhea (less than 3 loose stools/24 hours). Secondary objectives for Giardia infections are: 1) to compare the proportion of subjects with parasitological response (no detection of trophozoites on microscopic exam ) on Day 3, and 5; 2) to compare the rate of decrease of trophozoites/cyst load by qPCR in stools by Days 3 and 5; 3) to compare the proportion of subjects with negative stool antigens by days 3 and 5; 4) to compare the proportion of subjects with sustained cure (no detection of trophozoites by microscopic exam) at 14 and 28 days; 5) to compare the proportion of subjects with relapse (same strain) or re-infection (new strain) with positive stools at 14 and 28 days by genotyping the initial vs. subsequent strain; 6) to compare the time to resolution of diarrhea (less than 3 loose stools/24 hours).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Able to understand and comply with planned study procedures and be available for all study visits.
3. Male or non-pregnant non-lactating females 18-65 years of age, inclusive. Females of reproductive potential currently using effective contraceptive methods are eligible.
4. Amebiasis or giardiasis identified by rapid Enzyme Immunoassay (EIA) and positive antigen detection EIA of stool

   - if a subject is infected with both E. histolytica and Giardia, they will be enrolled in the E. histolytica study arm. Once the Entamoeba study arm is fully enrolled, any subsequent dual infected subjects will be enrolled in the Giardia arm. If a subject is infected with both Giardia and Cryptosporidium, they will not be enrolled.
5. Has diarrhea (defined as three or more loose stools) in the past 24 hrs, but is assessed to be clinically stable and in otherwise good health

   - as determined by medical history and targeted physical examination, if indicated based on medical history, to evaluate acute or currently ongoing chronic medical diagnoses or conditions that would affect the assessment of eligibility and safety of subjects. Existing medical diagnoses or conditions (except those in the Subject Exclusion Criteria) must be deemed as stable chronic medical conditions. A stable chronic medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last 3 months (90 days) and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months (180 days). Any change due to change of health care provider, insurance company, or that is done for financial reasons, as long as in the same class of medication, will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a violation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety. Topical, nasal, and inhaled medications, vitamins, and contraceptives are permitted.
6. Vital signs (oral temperature, pulse, and blood pressure) are all within normal protocol-defined ranges.
7. Laboratory tests (blood urea nitrogen, creatinine, aspartate transaminase (AST), alanine transaminase (ALT), white blood cells, platelets, and hemoglobin) are all within protocol-defined ranges. Subjects will be eligible for enrollment with the following laboratory values: blood urea nitrogen less than or equal to 30 mg/dL, creatinine less than or equal to 133 umol/L, AST or ALT less than or equal to 70.0 U/L, white cell count between 3.5 and 13.0 inclusive (10^9/L), platelets between 131 and 550 (10^9/L), hemoglobin between 11.0 and 18.0 gm/dL inclusive.
8. Urinalysis with no greater than trace protein. If a high protein is confirmed to be due to menstruation, it should be repeated.
9. Women of reproductive potential must have a negative urine pregnancy test within 72 hours of starting study medications.

   - Female subjects who are surgically sterile via tubal sterilization, bilateral oophorectomy or hysterectomy who have been postmenopausal for greater than 1 year are not considered to be of reproductive potential.
10. Female subjects participating in sexual activity that could lead to pregnancy must be using and continue to use highly effective contraception for a total of 4 months after enrollment.

    * Highly effective methods of contraception are defined as having low failure rates (i.e. less than 1 percent per year) when used consistently and correctly and may include, but are not limited to, abstinence from intercourse, monogamous relationship with a vasectomized partner, male condoms with spermicide, diaphragm with spermicide, intrauterine devices, and licensed hormonal methods. Females on effective forms of birth control will continue while on the study and for the follow-up period of 4 months total. The method and compliance of birth control used will be confirmed and documented at all study visits.

Exclusion Criteria:

1. Known intolerance of auranofin or gold compounds.
2. Pregnant or breastfeeding women or women of reproductive potential not using effective contraception or who plan to become pregnant or breastfeed at any given time during the study or within 3 months of study completion.
3. Use of metronidazole within the past 7 days.
4. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
5. Concurrent participation in other investigational protocols or receipt of an investigational product within the previous 30 days.
6. History of alcohol or drug abuse within the last five years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-11-06 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - International Center for Diarrheal Disease Research Bangladesh - Parasitology, Dhaka
  - Rajshahi Medical College Hospital, Rajshahi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were males and non-pregnant females between 18 to 65 years of age, inclusive, with amebiasis or giardiasis. Asymptomatic participants were recruited from the Mirpur community of Bangladesh by a randomized census. Symptomatic participants were identified by a health professional at either icddr,b or Rajshahi Medical College hospitals. Asymptomatic participants were enrolled from 06NOV2016 to 23APR2017. Symptomatic participants were enrolled from 16JAN2018 to 28JAN2021.
Groups:
- Asymptomatic E. Histolytica- Auranofin; Symptomatic E. Histolytica- Auranofin: 6mg auranofin daily x 7 days
  Auranofin: Auranofin is a gold-containing chemical salt available as 3mg capsules
- Asymptomatic E. Histolytica- Placebo; Symptomatic E. Histolytica- Placebo: 6mg placebo daily x 7 days
  Placebo: Placebo
- Asymptomatic Giardia- Auranofin; Symptomatic Giardia- Auranofin: 6mg auranofin daily x 5 days
  Auranofin: Auranofin is a gold-containing chemical salt available as 3mg capsules
- Asymptomatic Giardia- Placebo; Symptomatic Giardia- Placebo: 6mg placebo daily x 5 days
  Placebo: Placebo
Period: Overall Study
Arm/Group | Asymptomatic E. Histolytica- Auranofin | Asymptomatic E. Histolytica- Placebo | Asymptomatic Giardia- Auranofin | Asymptomatic Giardia- Placebo | Symptomatic E. Histolytica- Auranofin | Symptomatic E. Histolytica- Placebo | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo
Started | 0 | 1 | 17 | 16 | 0 | 0 | 30 | 29
Completed | 0 | 1 | 17 | 16 | 0 | 0 | 22 | 27
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
Not completed — COVID-19 Pandemic | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: No analyses performed on the following groups due to no participants enrolled: Asymptomatic E. histolytica- Auranofin, Symptomatic E. histolytica- Auranofin, Symptomatic E. histolytica- Placebo. Because only one participant was enrolled in Asymptomatic E. histolytica- Placebo, no analyses were performed.
Groups:
- Asymptomatic E. Histolytica- Placebo: 6mg placebo daily x 7 days
- Asymptomatic Giardia- Auranofin; Symptomatic Giardia- Auranofin: 6mg auranofin daily x 5 days
- Asymptomatic Giardia- Placebo; Symptomatic Giardia- Placebo: 6mg placebo daily x 5 days
- Total: Total of all reporting groups
Arm/Group | Asymptomatic E. Histolytica- Placebo | Asymptomatic Giardia- Auranofin | Asymptomatic Giardia- Placebo | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo | Total
Number analyzed (Participants) | 1 | 17 | 16 | 30 | 29 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 17 | 16 | 30 | 29 | 93
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (0) | 38.6 (9.3) | 33.5 (8.2) | 34.2 (9.5) | 33.4 (9.4) | 34.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 10 | 10 | 0 | 1 | 22
  Male | 0 | 7 | 6 | 30 | 28 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 17 | 16 | 30 | 29 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 17 | 16 | 30 | 29 | 93
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bangladesh | 1 | 17 | 16 | 30 | 29 | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Rapid Enzyme Immunoassay (EIA) and Positive Antigen Detection EIA for Giardia and Resolution of Diarrhea (Less Than 3 Loose Stools/24 Hours)
Description: Diarrhea was assessed by self-report at each study visit. Resolution of diarrhea occurred when participants reported less than 3 loose stools in 24 hours.
Time Frame: Day 5
Population: Modified Intention to Treat Population: All symptomatic participants who were randomized with available results, dispensed at least one dose of study medication, and had a positive rapid EIA and positive antigen detection EIA for Giardia at enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo
Number analyzed (Participants) | 29 | 29
Participants | 28 | 28
Statistical Analysis 1: Comparison: Symptomatic Giardia- Auranofin vs Symptomatic Giardia- Placebo; The null hypothesis is that the probability of resolution of diarrhea by Day 5 for participants receiving auranofin is equal to that for those receiving placebo; Test type: Superiority; p > 0.999, Fisher Exact — No adjustment for multiple comparisons was made. The a priori threshold for statistical significance is 0.05; Difference in Proportions = 0.00, 95% CI 2-sided [-0.12 to 0.12] — Adjusted Wald Intervals

2. Primary Outcome: Number of Participants With Positive Rapid Enzyme Immunoassay (EIA) and Positive Antigen Detection EIA for Giardia at Enrollment With Parasitological Response (no Detection of Cysts or Trophozoites on Microscopic Exam or Negative Antigen Test)
Description: Participants provided stool samples on Day 5. Stool samples were assessed for parasitological response by detection of cysts or trophozoites via microscopic exam or a negative antigen test.
Time Frame: Day 5
Population: Modified Intention to Treat Population: All asymptomatic participants who were randomized, dispensed at least one dose of study medication, and had a positive rapid EIA and positive antigen detection EIA for Giardia at enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Asymptomatic Giardia- Auranofin | Asymptomatic Giardia- Placebo
Number analyzed (Participants) | 14 | 14
Participants | 6 | 6
Statistical Analysis 1: Comparison: Asymptomatic Giardia- Auranofin vs Asymptomatic Giardia- Placebo; The null hypothesis is that the probability of parasitological response by Day 5 for participants receiving auranofin is equal to that for those receiving placebo; Test type: Superiority; p > 0.999, Fisher Exact — No adjustment for multiple comparisons was made. The a priori threshold for statistical significance is 0.05; Difference in Proportions = 0.00, 95% CI 2-sided [-0.34 to 0.34] — Adjusted Wald Intervals

3. Secondary Outcome: Proportion of Participants With Negative Giardia Stool Antigens
Description: Participants provided stool samples on Days 3 and 5. Stool samples were tested for Giardia using antigen detection EIA. Proportions are calculated as the number of participants with negative Giardia stool antigen tests divided by the number of participants with results available.
Time Frame: Day 3 through Day 5
Population: Modified Intention to Treat Population: All symptomatic participants who were randomized, dispensed at least one dose of study medication, had a positive rapid EIA and positive antigen detection EIA for Giardia at enrollment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo
Number analyzed (Participants) | 30 | 29
proportion of participants
  Day 3: number analyzed (Participants) | 29 | 29
  Day 3 | 0.45 [0.28 to 0.62] | 0.38 [0.23 to 0.56]
  Day 5: number analyzed (Participants) | 29 | 29
  Day 5 | 0.55 [0.38 to 0.72] | 0.34 [0.20 to 0.53]

4. Secondary Outcome: Proportion of Symptomatic Participants With Positive Rapid EIA and Positive Antigen Detection EIA for Giardia and Trophozoites on Smear at Enrollment With Parasitological Response
Description: Participants provided stool samples on Days 3 and 5. Stool samples were assessed for parasitological response by detection of trophozoites via microscopic exam. Proportions are calculated as the number of participants with parasitological response divided by the number of participants with results available.
Time Frame: Day 3 through Day 5
Population: Modified Intention to Treat Population: All symptomatic participants who were randomized, dispensed at least one dose of study medication, and had a positive rapid EIA and positive antigen detection EIA for Giardia at enrollment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo
Number analyzed (Participants) | 30 | 29
proportion of participants
  Day 3: number analyzed (Participants) | 29 | 29
  Day 3 | 0.97 [0.81 to 1.00] | 0.93 [0.77 to 0.99]
  Day 5: number analyzed (Participants) | 29 | 29
  Day 5 | 0.97 [0.81 to 1.00] | 1.00 [0.86 to 1.00]

5. Secondary Outcome: Proportion of Symptomatic Participants With Sustained Giardia Cure (no Detection of Trophozoites by Microscopic Exam)
Description: Participants provided stool samples on Days 14 and 28. Stool samples were assessed for sustained Giardia cure by detection of trophozoites via microscopic exam. Proportion is calculated as the number of participants with sustained cure divided by the number of participants with results available.
Time Frame: Day 14 through Day 28
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo
Number analyzed (Participants) | 30 | 29
proportion of participants
  Day 14: number analyzed (Participants) | 28 | 29
  Day 14 | 0.96 [0.81 to 1.00] | 0.90 [0.73 to 0.97]
  Day 28: number analyzed (Participants) | 24 | 28
  Day 28 | 0.96 [0.78 to 1.00] | 0.89 [0.72 to 0.97]

6. Secondary Outcome: Giardia Trophozoite/Cyst Load by Quantitative Polymerase Chain Reaction (qPCR) in Stools of Symptomatic Participants
Description: Participants provided stool samples on Days 3 and 5. The Giardia trophozoite/cyst load (parasites/uL) for each group was then assessed by Quantitative Polymerase Chain Reaction (qPCR).
Time Frame: Day 3 through Day 5
Population: Modified Intention to Treat Population: All symptomatic participants who were randomized, dispensed at least one dose of study medication, had a positive rapid EIA and positive antigen detection EIA for Giardia at enrollment, with available results.
Measure: Mean (95% Confidence Interval); unit: log parasite load/uL
Arm/Group | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo
Number analyzed (Participants) | 30 | 29
log parasite load/uL
  Day 3: number analyzed (Participants) | 28 | 28
  Day 3 | 8.6 [7.1 to 10.1] | 9.2 [8.0 to 10.4]
  Day 5: number analyzed (Participants) | 28 | 28
  Day 5 | 8.2 [6.8 to 9.6] | 8.1 [7.1 to 9.2]

7. Secondary Outcome: Time to Resolution of Diarrhea (Less Than 3 Loose Stools/24 Hours)
Description: as for outcome 1
Time Frame: Day 1 through Day 28
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo
Number analyzed (Participants) | 29 | 29
days | 3 [3.0 to 4.0] | 3 [NA to NA] — Not calculable due to low sample size and participants resolving at day 3.
Statistical Analysis 1: Comparison: Symptomatic Giardia- Auranofin vs Symptomatic Giardia- Placebo; The null hypothesis is that there is no difference in time to resolution of diarrhea between treatment arms, with a two-sided alternative; Test type: Superiority; p = 0.142, Log Rank — No adjustment for multiple comparisons was made. The a priori threshold for statistical significance is 0.05

8. Secondary Outcome: Proportion of Participants With Positive Rapid Enzyme Immunoassay (EIA) and Positive Antigen Detection EIA for Giardia at Enrollment With Parasitological Response (no Detection of Cysts or Trophozoites on Microscopic Exam or Negative Antigen Test)
Description: Participants provided stool samples on Day3. Stool samples were assessed for parasitological response by detection of cysts or trophozoites via microscopic exam or a negative antigen test. Proportions are calculated as the number of participants with parasitological response divided by the number of participants with results available.
Time Frame: Day 3
Population: Modified Intention to Treat Population: All participants who were randomized, dispensed at least one dose of study medication, and had a positive rapid EIA and positive antigen detection EIA for Giardia at enrollment.
Measure: Number (95% Confidence Interval); unit: proportion with parasitological response
Arm/Group | Asymptomatic Giardia- Auranofin | Asymptomatic Giardia- Placebo
Number analyzed (Participants) | 14 | 14
proportion with parasitological response | 0.43 [0.21 to 0.67] | 0.29 [0.11 to 0.55]

9. Secondary Outcome: Giardia Trophozoite/Cyst Load by Quantitative Polymerase Chain Reaction (qPCR) in Stools
Description: as for outcome 6
Time Frame: Day 3 through Day 5
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: log parasite load/uL
Arm/Group | Asymptomatic Giardia- Auranofin | Asymptomatic Giardia- Placebo
Number analyzed (Participants) | 14 | 14
log parasite load/uL
  Day 3 | 7.5 [5.0 to 10] | 9.0 [6.8 to 11.2]
  Day 5 | 7.1 [4.9 to 9.2] | 8.5 [6.3 to 10.8]

10. Secondary Outcome: Proportion of Asymptomatic Participants With Sustained Giardia Cure (no Detection of Trophozoites by Microscopic Exam)
Description: Participants provided stool samples on Days 14 and 28. Stool samples were assessed for sustained Giardia cure by detection of cysts or trophozoites via microscopic exam or negative antigen detection. Proportions are calculated as the number of participants with sustained cure divided by the number of participants with results available.
Time Frame: Day 14 through Day 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Asymptomatic Giardia- Auranofin | Asymptomatic Giardia- Placebo
Number analyzed (Participants) | 14 | 14
proportion of participants
  Day 14 | 0.29 [0.11 to 0.55] | 0.21 [0.07 to 0.48]
  Day 28 | 0.29 [0.11 to 0.55] | 0.14 [0.03 to 0.41]

11. Secondary Outcome: Proportion of Participants With Relapse (Same Strain) or Re-infection (New Strain) With Giardia-positive Stools by Genotyping the Initial vs. Subsequent Strain
Description: Participants provided stool samples on Days 14 and 28. Any stool that was still positive for Giardia or trophozoites at Days 14 and 28 had DNA genotyping of the parasite performed on de-identified specimens of extracted DNA. The genotypes from initial and final isolates were compared to determine relapse and/or re-infection. Proportion is calculated as the number of participants with relapse or re-infection divided by the number of participants with results available.
Time Frame: Day 14 through Day 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Asymptomatic Giardia- Auranofin | Asymptomatic Giardia- Placebo
Number analyzed (Participants) | 14 | 14
proportion of participants
  Day 14 - Relapse: number analyzed (Participants) | 12 | 12
  Day 14 - Relapse | 0.58 [0.32 to 0.81] | 0.75 [0.46 to 0.92]
  Day 14 - Re-infection: number analyzed (Participants) | 12 | 12
  Day 14 - Re-infection | 0.33 [0.14 to 0.61] | 0.25 [0.08 to 0.54]
  Day 28 - Relapse: number analyzed (Participants) | 8 | 11
  Day 28 - Relapse | 0.63 [0.30 to 0.87] | 0.73 [0.43 to 0.91]
  Day 28 - Re-infection: number analyzed (Participants) | 8 | 11
  Day 28 - Re-infection | 0.25 [0.06 to 0.60] | 0.09 [0.00 to 0.40]

12. Secondary Outcome: Proportion of Participants With Relapse (Same Strain) or Re-infection (New Strain) With Giardia-positive Stools by Genotyping the Initial vs. Subsequent Strain
Description: Participants provided stool samples on Days 1, 14 and 28. Participants that were positive for Giardia via antigen detection at Day 1 and had a negative antigen detection test followed by a positive antigen detection test had DNA genotyping of the parasite performed on de-identified specimens of extracted DNA. The genotypes from initial (Day 1) and final isolates (Day 14/28) were compared to determine relapse and/or re-infection. Proportion is calculated as the number of participants with relapse or re-infection divided by the number of participants with results available.
Time Frame: Day 1 through Day 28
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo
Number analyzed (Participants) | 30 | 29
proportion of participants
  Day 14 - Relapse: number analyzed (Participants) | 12 | 15
  Day 14 - Relapse | 0.08 [0.00 to 0.38] | 0.07 [0.00 to 0.32]
  Day 14 - Re-infection: number analyzed (Participants) | 12 | 15
  Day 14 - Re-infection | 0.00 [0.00 to 0.28] | 0.07 [0.00 to 0.32]
  Day 28 - Relapse: number analyzed (Participants) | 9 | 14
  Day 28 - Relapse | 0.11 [0.00 to 0.46] | 0.07 [0.00 to 0.34]
  Day 28 - Re-infection: number analyzed (Participants) | 9 | 14
  Day 28 - Re-infection | 0.00 [0.00 to 0.34] | 0.14 [0.03 to 0.41]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the participants received study product and continued through study day 29.
Description: Adverse events were collected at each visit using specific questions and/or targeted physical examination. No adverse events were collected for the following groups due to no participants enrolled: Asymptomatic E. histolytica- Auranofin, Symptomatic E. histolytica- Auranofin, Symptomatic E. histolytica- Placebo.
Arm/Group | Asymptomatic E. Histolytica- Placebo | Asymptomatic Giardia- Auranofin | Asymptomatic Giardia- Placebo | Symptomatic Giardia- Auranofin | Symptomatic Giardia- Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/17 | 0/16 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/17 | 0/16 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/1 | 9/17 | 7/16 | 0/30 | 2/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asymptomatic E. Histolytica- Placebo (N=1) | Asymptomatic Giardia- Auranofin (N=17) | Asymptomatic Giardia- Placebo (N=16) | Symptomatic Giardia- Auranofin (N=30) | Symptomatic Giardia- Placebo (N=29)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess Rupture (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT02736968/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT02736968/SAP_001.pdf